CLINICAL TRIAL: NCT03487991
Title: Stress, Sleep and Cardiovascular Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Howard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL136626-01 (NIH)
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Posttraumatic Stress Disorder; Insomnia
Keywords: autonomic balance; sleep; endothelial function; behavior; stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- personalized behavioral recommendations (Experimental): Will receive recommendations for altering sleep related behavior based on data from in-home monitoring.
  Interventions: Behavioral: Personalized sleep intervention
- educational control (No Intervention): Will receive the data without recommendations. Will receive personalized recommendations after the follow up assessment.

INTERVENTIONS:
Behavioral: Personalized sleep intervention — Personalized feedback and recommendations based on study observations of sleep behavior and how participants cope with potentially sleep disruptive cognitions on their frequency and impact and on sleep efficiency. A written report is provided to participants and their initial modifications are monitored.
  Arms: personalized behavioral recommendations

SUMMARY:
We are evaluating a model where trauma exposure and threatening environments elicit nocturnal vigilance and sleep-related fears that compromise the healthy reduction of autonomic arousal during sleep which in turn stimulates secretion of atherogenic humoral factors, arterial stiffening, and cardiovascular disease risk. We will examine the roles of pre-sleep cognition using a questionnaire and real time assessment, and modifiable strategies for coping with sleep disruptive cognitions. We will then evaluate the impact of providing personalized feedback and recommendations based on study observations on how participants cope with potentially sleep disruptive cognitions and sleep efficiency in a randomized trial.

DETAILED DESCRIPTION:
The study has 3 specific aims.

Aim 1. To confirm the effects of neighborhood and posttraumatic stress, and nocturnal vigilance on nocturnal autonomic balance determined by complementary biomarkers.

Hypothesis 1a - Neighborhood disorder and posttraumatic stress symptom severity will be inversely correlated with indicators of autonomic balance derived from analyses of heart rate variability and cardiac impedence, and nocturnal/evening urinary noradrenergic excretion ratios.

Hypothesis 1b - These relationships will be partially or fully accounted for by nocturnal vigilance and the frequency and intensity of pre-sleep disruptive cognitions assessed in real time, and strategies for coping with sleep disruptive thoughts.

Aim 2. To determine relationships of nocturnal autonomic activity to biomarkers of inflammation and endothelial dysfunction.

Hypothesis 2 - Indicators of nocturnal autonomic balance will correlate with morning levels of pro-inflammatory cytokines and adhesion molecules; and pulse wave velocity.

Aim 3. To determine if sleep is improved 6 months after receiving personalized recommendations for adaptively modifying sleep-related behaviors, and if improved sleep and reduced pre-sleep cognitive arousal are associated with more favorable nocturnal autonomic balance and endothelial function.

Hypothesis 3a - Reduced frequency and intensity of sleep disruptive cognitions and improved sleep efficiency will be more likely in the group that received personalized feedback and recommendations for sleep.

Hypothesis 3b - Reduction of disruptive pre-sleep cognitions, and increased sleep efficiency will be associated with improved autonomic status at night and a more favorable profile of cardiovascular risk biomarkers.

ELIGIBILITY:
Inclusion Criteria:1. Healthy adults age 18 - 35, self-identified as Black or African American, born in the United States.

Exclusion Criteria:

* current medical or psychiatric condition that affects sleep or requires daily - use of medication other than PTSD, phobic disorders, or past history of major depression
* severe alcohol or drug use disorders
* overnight shift worker or an extreme chronotype
* sleep disorder other than insomnia or nightmares
* morbid obesity (body mass index > 40)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
sleep efficiency | 6 months
  percent of time in bed spent asleep

SECONDARY OUTCOMES:
normalized high frequency ratio of heart rate variability while in bed | 6 months
  an index of parasympathetic nervous system activity
pulse wave velocity | 6 months
  a measure of arterial elasticity

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Unit; Howard University Hospital, Washington D.C., District of Columbia, United States